CLINICAL TRIAL: NCT05228106
Title: Pragmatic Study on the Use of 68Ga-PSMA-617 PET/CT Imaging as a Standard of Care to Influence Clinical Management of Tumors Overexpressing PSMA.
Brief Title: 68Ga-PSMA-617 PET/CT for PSMA-expressing Tumor: a Pragmatic Study
Status: Recruiting | Type: Observational
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: PSMA-2022-4331
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Solid Cancers
Keywords: [68Ga]-PSMA-617; PET imaging; Pragmatic study; PSMA-expressing cancers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients eligible for [68Ga]-PSMA-617-PET: All cancer patients referred by their physician and fulfilling the eligibility criteria across Canada can be recruited to the primary site of the study. Patients will be injected intravenously with a [68Ga]-PSMA-617 dose calculated depending on the characteristics of the PET tomograph and patient weight (maximum 370 MBq). 60-90 minutes following injection, patients will be imaged in a PET/CT scanner. Images will be analyzed by a trained nuclear medicine physician. Safety profile, eventual adverse effects, false positives, false negatives and any abnormal biodistribution of the radiotracer will be monitored and analysed.
  Interventions: Diagnostic Test: [68Ga]-PSMA-617

INTERVENTIONS:
Diagnostic Test: [68Ga]-PSMA-617 — The intervention consists of an intravenous injection of the radiopharmaceutical [68Ga]-PSMA-617 and a physiological saline flush, followed 60-90 minutes later by a PET/CT image acquisition.
  Other Names: PSMA-PET

SUMMARY:
This project aims to monitor the innocuity/safety profile of cyclotron-produced [68Ga]-PSMA-617 PET imaging in PSMA-expressing cancers. It is a single-site, pragmatic, non-randomized and open-label study, with no control group. Although prostate cancers constitute the usual recommended population for this PET modality, recent evidences suggest that most solid tumors express substantial amount of PSMA in their neovasculature. As such, all cancers (excluding non-solid cancers) will be eligible for [68Ga]-PSMA-617 PET imaging in this trial, for as long as their tumors express PSMA.

This study also aims to instigate the use of [68Ga]-PSMA-617 in the routine standard-of-care for detection and follow-up of eligible cancers. FInally, this project seeks to gather information about the impact on patient management this novel PET modality will have over the current standard-of-care.

DETAILED DESCRIPTION:
In developed countries such as Canada, prostate cancers are the most frequently diagnosed and the third deadliest cancer among men. Early detection and management of low-stage prostate cancer leads to a 5-year survival rate nearing 100%. However, advanced and metastatic prostate cancers remain a clinical challenge to both assess and treat, despite significant advances in the field in the last years.

Among the best existing diagnostic tools for advanced cancers overall, FDG-PET suffers from a very low sensitivity for prostate cancers. Indeed, not only those lesions are most of the time hypometabolic and indolent, but also loco regional assessment is heavily impaired by the proximity of the background-generating, radio metabolite-rich bladder. Other imaging modalities such as Computed Tomography (CT) and Magnetic Resonance imaging (MRI) do not perform better, and are also plagued with relatively low sensitivity and specificity. As such, alternative, PET tracers were developed in order to better assess metastatic prostate cancers. One of the earliest attempts was with choline-derived tracers (either labeled with 11C or 18F) which showed superior diagnostic properties than FDG, but still harbors a range of sensitivity from poor to excellent depending of the site of the lesions. Recently, the amino acid analog 18F-fluciclovine (Axumin) showed great promises thanks to a low renal excretion and high prostate tumor uptake which resulted in much improved sensitivity. However, while both choline and fluciclovine offer precise prostate cancer diagnostic, they do not provide much information about the prognostic of the disease or the efficacy of targeted therapies.

The Prostate Specific Membrane Antigen (PSMA) is a transmembrane glycoprotein with folate hydroxylase and glutamate carboxypeptidase enzymatic activities. PSMA was first reported to be strongly expressed in more than 90% of prostate cancers. Moreover, PSMA expression on prostate tumors is proportional to the plasmatic concentration of the routinely-assessed Prostate Specific Antigen (PSA), which is currently the main screening and treatment follow-up tool for prostate cancer. PSMA overexpression occurs most frequently in high-grade and metastatic diseases, as well as for castration-resistant cancers. As such, PSMA constitutes a target of choice for an imaging modality aiming for prognosis and treatment assessment of prostate cancers, as well as for targeted endoradiotherapy.

High PSMA expression was also observed in the neovasculature of most solid tumors, notably breast, lung and gastrointestinal cancers. 68Ga-PSMA-PET was reported to allow high-uptake detection of nonprostate cancers. More recently, a preliminary clinical report showed that breast cancers can readily be imaged using 68Ga-PSMA, with the highest detection rate observed in the triple-negative subtype. As such, while 68Ga-PSMA was mainly explored in prostate cancers until now, rising evidence demonstrates its applicability to most solid cancers as well.

In the last few years, many peptidomimetic compounds were designed as PSMA-specific ligands, such as PSMA-11, PSMA-617 and PSMA-1007. The latter is radiolabeled covalently with a 18F, whereas most other molecules depend upon their chelator moiety for labeling with a radiometal such as 64Cu or 68Ga. The main advantages of using a chelator-bearing compound include ease of labeling and purification along with the potential to alternatively label with therapeutic radiometals such as 177Lu or 225Ac to form a theranostic pair with PET-capable isotopes with the same molecular frame. Notably, PSMA-617, labeled with 68Ga for PET imaging and with 225Ac for therapy, showed astonishing potential in a cohort of advanced prostate cancer.

The current trial aim to investigate the use of cyclotron-produced 68Ga chelated in PSMA-617 for the diagnostic, prognostic and treatment follow-up of PSMA-overexpressing cancers. The relative performances and safety profile of the cyclotron-produced 68Ga-PSMA-617 at our center with the available clinical data from the literature. Moreover, the sensitivity, specificity and diagnostic performance of 68Ga-PSMA-617 will be compared with the current standard of care for PSMA+ cancer diagnostic and follow-up.

TUMORS THAT MAY BE VISUALIZED WITH 68GA-PSMA-617 PET/CT The sensitivity of 68Ga-PSMA-617 PET/ CT is likely to vary among tumor grade, PSA blood levels and depending on the density of PSMA in the tumors. PSMA is expressed by healthy prostate tissue, but at a baseline level compared to the overexpression assessed in prostate cancers. High PSMA levels were also reported in most glioma, lung, gastrointestinal, liver, breast, pancreatic and thyroid cancers, among others. As such, 68Ga-PSMA-617 is expected to enable precise detection and follow-up for all those indications.

High uptake is expected in the salivary glands; such foci should not be confounded with tumor lesions.

CLINICAL USES

In the management of cancers overexpressing PSMA, 68Ga-PSMA-617 PET/CT is recommended or under investigation for the following:

* Disease staging
* Follow-up of patients with known disease to detect residual, recurrent, or progressive disease (restaging)
* Determine PSMA status visually as well by using semi-quantitative parameters like standardized uptake value (SUV)
* Monitoring response to therapy

ELIMINATION ROUTE 68Ga-PSMA-617 is rapidly cleared from the blood. Arterial elimination of activity is bi-exponential, and no radioactive metabolites are detected after 12h in the serum or urine. 68Ga-PSMA-617 tumor uptake increases steadily through time. Excretion occurs via both the urinary and the hepatobiliary pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical requisition for a 68Ga-PSMA-617 PET/CT signed by a referring doctor;
2. Patients with suspected, proven or prior tumor expressing PSMA;
3. Informed consent by patient.

Exclusion Criteria:

1. Patient refusal to participate;
2. Prior severe anaphylactic reaction to 68Ga-PSMA-617 .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study will recruit all eligible patients referred to our center for PET/CT imaging with [68Ga]-PSMA-617 for 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) of 68Ga-PSMA-617 | 5 years
  Following the injection, the patient will be explicitly reminded of possible symptoms and undesirable events. The patient will be advised to inform the study personnel of the occurrence of any events, at the most opportune time. The patient will be instructed to call the local nuclear medicine study coordinator for any undesirable event that may occur for 48 hours after the PET/CT scan.
  Safety will be assessed by compiling all reported adverse events. Adverse events reported by patients or observed by the investigator will be recorded in the patients' CRFs, the AE database, and reported to the research manager.

SECONDARY OUTCOMES:
Generate clinical information on the impact of [68Ga]-PSMA-617 for cancer patient management | 5 years
  PSMA-PET is routinely used to assess and follow-up prostate cancers with unprecedented precision. Recent reports found that most solid cancers are also susceptible to be detected and managed with this modality. This trial offers the opportunity to evaluate the impact of this state-of-the-art diagnostic procedure on the management of eligible cancers patients on a large, nation-wide cohort.
Instigate the routine standard-of-care use of [68Ga]-PSMA-617 for eligible cancer patients | 5 years
  Clinical and scientific evidences hinted that [68Ga]-PSMA-617 might be a complementary, even superior diagnostic tool than the current standard-of-care FDG-PET/CT for solid tumors. As such, this trial aims to implement [68Ga]-PSMA-617 as the new standard-of-care for precision diagnostic of NETs.

CONTACTS AND LOCATIONS:
Overall Officials: Éric E Turcotte, MD, Principal Investigator — Université de Sherbrooke, Centre de Recherche du CHUS
Locations (1):
- CHUS, Sherbrooke, Quebec, Canada